CLINICAL TRIAL: NCT03881787
Title: Clinical Trial to Evaluate Pharmacokinetics,Safety and Immunogenicity of Single Injection of Recombinant Anti-EGFR Human Mouse Chimeric Monoclonal Antibody Injection (CDP1) to Healthy Volunteers Compared to Erbitux
Brief Title: Clinical Trial to Evaluate Pharmacokinetics,Safety and Immunogenicity of Single Injection of CDP1 to Healthy Volunteers Compared to Erbitux
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dragonboat Biopharmaceutical Company Limited (Industry)
Collaborators: West China Hospital (Other); Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDP100002
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-EGFR monoclonal antibody (Experimental): Recombinant anti-EGFR human mouse chimeric monoclonal antibody injection 250mg/m2 single administration
  Interventions: Drug: anti-EGFR monoclonal antibody
- Cetuximab (Active Comparator): Cetuximab,Erbitux 250mg/m2 single administration
  Interventions: Drug: Cetuximab injection

INTERVENTIONS:
Drug: anti-EGFR monoclonal antibody — Recombinant anti-EGFR human mouse chimeric monoclonal antibody injection
  Other Names: CDP1
  Arms: anti-EGFR monoclonal antibody
Drug: Cetuximab injection — Cetuximab injection
  Other Names: Erbitux
  Arms: Cetuximab

SUMMARY:
Background Colorectal cancer (CRC) is one of the most common human malignant tumors. The incidence and mortality of colorectal cancer in our country are on the rise. Surgery-based, combined with chemotherapy, radiotherapy comprehensive treatment, is the main treatment of colorectal cancer. Surgical resection has been recognized as the primary treatment of colorectal cancer. However, due to the majority of patients already advanced at the time of diagnosis, some difficulties are brought to radical surgery. Therefore, the importance of chemotherapy for colorectal cancer gradually been clinically recognized, But rarely survive more than 18 months." In addition to chemotherapy, there is now a more ideal model of cancer treatment- molecular targeted therapies, including monoclonal antibody drugs such as cetuximab, as well as small molecule tyrosine kinases Inhibitors gefitinib and so on. Molecular targeted drugs make use of the difference in molecular biology between tumor cells and normal cells. Targeting drugs to tumor cells and inhibiting the growth and proliferation of the cells can achieve the therapeutic effect, which has the advantages of high specificity and low adverse reaction. The bio-targeted drug cetuximab is the first drug approved to marketed as an epidermal growth factor receptor (EGFR)-targeting immunoglobulin 1（IgG1）monoclonal antibody. Cetuximab, either monotherapy or combined radiotherapy and chemotherapy, can exert excellent anti-tumor activity in EGFR-positive malignant tumors and can significantly enhance the efficacy of radiotherapy and chemotherapy.

Reference to cetuximab injection, guilin sanjin Co., Ltd. and dragonboat Co., Ltd. jointly developed a recombinant anti-EGFR human mouse chimeric monoclonal antibody (R & D code: CDP1).The primary structure of CDP1 is exactly the same with cetuximab, the higher structure and Physical and chemical properties and cetuximab are highly similar. Pharmacodynamic activity in vivo and in vitro, pharmacokinetic characteristics and toxicological reactions are also similar to cetuximab. CDP1 selected with cetuximab consistent formulations, prescriptions, specifications.

CDP1 was approved by China Food and Drug Administration (No. 2016L06884) in August 2016 for clinical studies. According to the contents of the document and guidelines for biological analogs, the clinical pharmacokinetic and clinical effectiveness comparison tests of CDP1 and the safety and immunogenicity assessment are planned.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

To compare the pharmacokinetic characteristics of a single dose between CDP1 and the original drug Erbitux in healthy volunteers.

Secondary :

To compare the safety and immunogenic characteristics of the single dose between CDP1 and the original drug Erbitux in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers participate in clinical trials voluntarily and sign informed consent.
2. Age 18 ~ 45 (inclusive) years , male.
3. The body weight is not less than 50 kg, and the body mass index is between 18.5 and 26 (including both ends).
4. Good health, no heart, liver, kidney or other acute or chronic digestive tract diseases, respiratory diseases, blood, endocrine, nervous, mental and other systemic diseases.
5. Physical examination, vital signs, blood routine, urine routine, blood biochemistry, electrocardiogram and chest X-ray examination are all normal, or the abnormal results of the examination are not clinically meaningful by the investigator.
6. Agree to avoid spouse pregnancy during the trial period and within 6 months after the end of the administration.

Exclusion Criteria:

1. Allergic constitution, those who are allergic to the test drug ingredients or have a history of allergies to any drug or food or a history of pollen allergy; those with abnormal serum immunoglobulin E (IgE) (more than 3 times higher than the upper limit of normal).
2. Anti-drug antibody (ADA) positive.
3. Infections currently in need of clinical treatment.
4. HBsAg, HBeAg, HCV-Ab, HIV-Ab or TP-Ab positive.
5. Upon inquiry, there is a clear current medical history of the central nervous system, cardiovascular system, kidney, liver, digestive system, respiratory system, metabolic system or other significant diseases.
6. Upon inquiry, a person with a history of mental illness.
7. Upon inquiry, there is a history of cancer and it is judged by the investigator that it is not suitable for participation.
8. According to the investigator's judgment, the investigator believes that it is not suitable for the participants in this clinical trial for various reasons.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters: Area Under the Serum Concentration-time Curve From Time Zero to the Last Sampling Time (AUC0-t) After Infusion | Up to 22 Days
  AUC(0-t) for CDP1

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUC0-00) After Infusion | Up to 22 Days
  Pharmacokinetic parameters: AUC(0-00) for CDP1
Pharmacokinetic parameters: Observed Maximum Serum Concentration (Cmax) of CDP1 After Infusion | Up to 22 Days
  Pharmacokinetic parameters Cmax for CDP1
Pharmacokinetic parameters: Mean Residence Time of Drug in the Body (MRT) of CDP1 After Infusion | Up to 22 Days
  Pharmacokinetic parameters MRT for CDP1
Pharmacokinetic parameters: Apparent Terminal Half-life (t1/2) of CDP1 After Infusion | Up to 22 Days
  Pharmacokinetic parameters T1/2 for CDP1
Pharmacokinetic parameters: Total Body Clearance of Drug From Serum (CL) After Infusion | Up to 22 Days
  Pharmacokinetic parameters CL for CDP1
Vital signs: Blood pressure | Up to 29 Days
  Vital signs: Blood pressure
Vital signs: Pulse rate | Up to 29 Days
  Vital signs: Pulse rate
Vital signs: Respiratory rate | Up to 29 Days
  Vital signs: Respiratory rate
Physical examination: Weigh | Up to 29 Days
  Physical examination: Weigh
Frequency of adverse events (AE) | Up to 29 Days
  Frequency of adverse events (AE)
Immunogenicity indicators: Anti-drug antibodies (ADA) | Up to 29 Days
  Immunogenicity indicators: Anti-drug antibodies (ADA)
Immunogenicity indicators: neutralizing antibodies | Up to 29 Days
  Immunogenicity indicators: neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: zheng li, doctor, Principal Investigator — West China Hospital; zhu tongyu, doctor, Study Director — Shanghai Public Health Clinical Center
Locations (2):
- China (2):
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuang